CLINICAL TRIAL: NCT07345975
Title: Characterization of Opposition to Organ Donation at Strasbourg University Hospital in 2024-2025
Acronym: OPPO-PMO
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9824
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Organ Donation
Keywords: Organ Donation; Organ transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In 2024, 29,000 people are waiting for organ transplants in France, and only 6,034 transplants were performed during the year. 852 people died while waiting for a transplant. The gap between the number of available transplants and the number of patients waiting for transplants has been widening since the 1990s; there is talk of a shortage of transplants. There is therefore an urgent need to find more transplants and mobilize the entire population to this end.

French law supports presumed consent, meaning that we are all donors unless we have expressed otherwise during our lifetime. In fact, 80% of French people say they are in favor of organ donation after their death, but few discuss it with their loved ones. When families are approached about multi-organ removal to gather any opposition from the deceased, the refusal rate is 37% (compared to an expected 20%).

It is difficult to determine whether this opposition truly comes from the deceased themselves, their loved ones, uncertainty, or the situation. As this is the leading cause of non-donation, it is essential to better characterize this opposition in order to reduce it and allow for more organ donation and, ultimately, transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are brain dead and/or eligible for a Maastricht 3 protocol (discontinuation of active treatment with death due to circulatory arrest in intensive care)
* Hospitalized in the intensive care unit of the Strasbourg University Hospital or transferable to the Strasbourg University Hospital for multi-organ removal (anticipated approach)
* Existence of relatives with whom discussion is possible
* Presence of organ procurement coordination at the initial donation interview

Exclusion Criteria:

* Absence of relatives of the deceased (no interview with them)
* Absence of organ procurement coordination during the initial discussion with relatives regarding organ and tissue procurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are brain dead and/or eligible for a Maastricht 3 protocol (discontinuation of active treatment with death due to circulatory arrest in intensive care)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-14 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02-14 (Estimated)

PRIMARY OUTCOMES:
Distribution of positions regarding organ donation (certain, uncertain, unknown) | Up to 12 months
  Distribution of positions regarding organ donation (certain, uncertain, unknown):
  For illustration purposes:
  * Certain position: ≈ 65%
    * Favorable: ≈ 55%
    * Opposed: ≈ 10%
  * Uncertain position: ≈ 25%
  * Unknown/unexpressed position: ≈ 10%

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie, Réanimation et Médecine Périopératoire - CHU de Strasbourg - France, Strasbourg, France